CLINICAL TRIAL: NCT04361773
Title: Effect of Photobiomodulation on the Treatment of Soft Tissue Traumatic Injuries: Study Protocol for a Double-Blind, Randomized, Controlled Trial
Brief Title: Effect of Photobiomodulation on the Treatment of Soft Tissue Traumatic Injuries
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TraumaSoftTissue
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Soft Tissue Injuries
MeSH Terms: conditions — Soft Tissue Injuries | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Researchers who will carry out the application of PBM will not carry out any type of evaluation. The evaluations (initial and after application of the FBM) will be made by the field researchers, who will not be informed of the group in which each participant is allocated. Participants will not be aware of whether or not they have received PBM, as the applicator researchers will position the equipment at the irradiation sites in all participants, cover the limb with fabric that does not allow visualization, and will only activate the light when and where provided in the specific experimental group. A sound recorded on a cell phone will be played when the participant is allocated to the sham group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation group (Active Comparator): In this group, PBM will be applied daily using LED devices until the lesion presents healthy granulation tissue, absence of necrosis and purulent secretion and, therefore, is suitable for primary closure, closure by flap or graft or for healing by second intention. At this point, the protocol will be finalized.
  Interventions: Radiation: Photobiomodulation
- Sham group (Sham Comparator): Sham group participants will receive the application of the disconnected device, for the same period. The characteristic sound of the device will be activated by means of recording.
  Interventions: Other: Sham Photobiomodulation

INTERVENTIONS:
Radiation: Photobiomodulation — Treatment with a device with 144 light emitting diodes (LEDs) at wavelengths of 420, 660 and 850nm, 3J per point for 10 minutes.
  Arms: Photobiomodulation group
Other: Sham Photobiomodulation — Simulation of the LED application, with a device with external characteristics identical to that of the PBM group, for the same period of time.
  Arms: Sham group

SUMMARY:
Soft tissue injuries are directly related to the energy of the trauma and its repair is the main factor for bone healing and the recovery of the function of the affected limb. Photobiomodulation (PBM) is indicated as an adjuvant treatment to accelerate wound healing, however, there is still a lack of evidence regarding its effect on traumatic soft tissue injuries. This project aims to evaluate the effects of the application of PBM in the resolution of complex soft tissue injuries of traumatic origin associated with tibial fractures. 84 adult individuals, aged between 18 and 60 years, hospitalized with tibial fractures awaiting resolution of soft tissue injuries will be included to undergo definitive surgery. The subjects will be randomized in two groups: PBM (treated with a device with 144 LED emitting diodes at wavelengths of 420, 660 and 850nm, 3J per point for 10 minutes) and Sham (simulation of the LED application, with a device with characteristics identical to that of the PBM group, for the same period of time). Subjects will be treated daily until release for surgery. The primary outcome will be the assessment of the wound healing process using the BATES-JENSEN scale. Secondary outcomes will be: pain intensity; consumption of analgesic drugs; serum evolution of inflammatory markers C-reactive protein and creatine kinase, measurement of the lesion area, time needed for release for definitive surgery, presence of infection, and the cost-effectiveness of PBM. The evaluations will be carried out before the beginning of the intervention and daily until the participant is considered ready for surgery (which will be considered the end of the experimental period). Data will be analyzed statistically considering a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals of both sexes, aged between 18 and 60 years;
* Interned in the Orthopedics and Infirmary Emergency Room of the Surgical Clinic of Conjunto Hospitalar do Mandaqui;
* Victims of high-energy trauma in the lower limbs with sufficient soft tissue injury to make primary closure unfeasible or definitive treatment of injuries in the initial care associated with tibial fracture.

Exclusion Criteria:

* Diagnosis of chronic systemic diseases (renal failure, diabetes mellitus, hypertension, peripheral vascular insufficiency);
* Allergy to cefazolin and gentamicin;
* Uncontrollable active bleeding;
* Occlusive arteriopathies;
* Compartmental syndrome;
* Necrosis in the area of neurovascular injury with sensory deficit at the injury site;
* History of previous surgeries on the affected limb;
* Local or systemic changes that contraindicate surgical intervention or hinder the postoperative period;
* Smoking;
* Photo sensitivity history;
* Neurological and psychiatric disorders;
* Use of anti-inflammatory drugs in the last 15 days prior to the trauma;
* Pregnant women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-05-30 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of the wound healing process using the BATES-JENSEN scale | Baseline and through study completion, an average of 1 month.
  Evaluation of the healing process of soft tissue injuries in lower limbs associated with tibial fractures caused by high-energy trauma using the variation in the Bates Jensen Wound Assessment Tool scale score. The current version of BWAT contains 13 items that measure size, depth, borders, detachment, type and amount of necrotic tissue, type and amount of exudate, edema and hardening of the peripheral tissue, skin color around the wound, granulation tissue and epithelialization. The measurement scale is of the Likert type, with five points, where 1 indicates the best condition of the wound and 5, the worst condition. The total score is obtained with the sum of all items and can vary from 13 to 65 points, with the highest scores indicating the worst wound conditions. The items size, depth, edges and detachment should be scored as zero when the lesions are healed. The instrument contains two additional items - location and shape - that are not part of the total score.

SECONDARY OUTCOMES:
Change in Pain Intensity Through VAS | Baseline and through study completion, an average of 1 month.
  Pain will be assessed by field researchers by applying the visual analogue pain scale (VAS). This scale is represented by a 10 cm line, with the phrases "no pain" and "unbearable pain" at its ends.
Consumption of painkillers | Baseline and through study completion, an average of 1 month.
  The type, dosage and frequency of analgesic consumption will be checked and recorded daily during the medical visit by the field team responsible for the daily medical visit. The results will be passed on to the main researcher for storage, tabulation and interpretation.
Change in serum evolution of inflammatory markers | Baseline, every three days and through study completion, an average of 1 month.
  For laboratory evaluation of the evolution of the inflammatory process and muscle damage, the following tests will be collected: C-reactive protein (CRP), Creatinophosphokinase (CPK), serum urea, creatinine, blood count and coagulogram. These exams will be collected at the time of admission, every three days and when the soft parts are resolved.
Change in Lesion Area Measurement | Baseline and through study completion, an average of 1 month.
  The wounds will be photographed along with a cut of graph paper using the camera of the iPhone 8 mobile device, to allow the calibration of the measurement application. The photos will be taken by the doctors who will visit the patient daily at the patient's bed and pass them on to the main researcher. The images will be stored and later evaluated with the aid of the Image J® application, a public domain Java image processor and analyzer, developed by Wayne Rasband of the Research Services Branch, National Institute of Mental Health, Bethesda, Maryland.
Time needed for liberation for definitive surgery | Baseline and through study completion, an average of 1 month.
  Each lesion will be considered solved when it presents healthy granulation tissue, without necrosis or purulent secretion and is, therefore, suitable for primary closure, flap or graft closure or apt to choose healing by second intention. At this point, the protocol will be finalized and this data will be added to the study participant's medical record.
Presence of Infection | Baseline and through study completion, an average of 1 month.
  Field researchers will collect information regarding the patient's temperature, blood pressure and heart rate every 24 hours. In addition, the wound will be evaluated for the presence of secretion, necrosis, odor and color. If the wound shows signs of infection (purulent secretion, foul odor, areas of superficial or deep necrosis, accompanied or not by systemic signs such as fever, a fall in general condition, lack of appetite), surgical cleaning of the wound will be indicated, and at this moment, collections of samples for culture and photographs before and after surgical debridement will be carried out by field researchers. The patient will be excluded from the study.
Cost effectiveness of Photobiomodulation | Baseline and through study completion, an average of 1 month.
  The cost-effectiveness establishes whether or not a treatment should be implemented as a therapeutic measure, being calculated by the difference between the cost of two interventions proposed as treatment divided by the difference between its consequences. For the evaluation of the cost-effectiveness of photobiomodulation, the "reduction in the score of the Bates Jensen scale" will be considered as the outcome.
Change in Peripheral Perfusion through Clinical Evaluation | Baseline and through study completion, an average of 1 month.
  The peripheral perfusion of the affected limb will also be evaluated clinically by two doctors, through palpation of the distal pulses (pedicle and posterior tibial), pain and passive extension of the fingers (to clinically assess the occurrence of compartment syndrome) capillary filling time, limb, granulation of the wound, occurrence of superficial or deep necrosis. In case of vascular involvement of the limb, joint assessment with the vascular surgery service will be requested and the case will be excluded from the study.